CLINICAL TRIAL: NCT03304938
Title: Efficacy and Safety of Lavender Aromatherapy on Sleep Quality and Metabolic Parameters of Type 2 Diabetic Patients With Insomnia
Brief Title: Lavender Aromatherapy on Sleep Quality and Metabolic Parameters of Type 2 Diabetic Patients With Insomnia
Acronym: LavenAromDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of internal medicine and endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 95010112052
Record Dates: First submitted 2017-07-25; First posted 2017-10-09 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 2; Sleep Disturbance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Parasomnias | interventions — lavender oil

STUDY DESIGN:
Intervention Model Description: 40 diabetic patients with sleep disorder with the inclusion criteria will enter into the crossover study and randomly assign to treatment or placebo groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Lavender Essential oil as medication and almond oil as placebo put in similar dark buttle and the head of placebo bottle aromatized whit Lavender Essential oil and all of participants, care provider, investigator and outcomes assessor will be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender oil (Active Comparator)
  Interventions: Drug: Lavender Oil
- vehicle (Almond oil) (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Lavender Oil — The intervention group pour 3 drops of Lavender essential oil on a cotton wool then smell it rhythmic and slowly for 5 minutes at bed time for 4 weeks
  Arms: Lavender oil
Drug: Placebos — The placebo group pour 3 drops of Almond oil on a cotton wool then smell it rhythmic and slowly for 5 minutes at bed time for 4 weeks
  Arms: vehicle (Almond oil)

SUMMARY:
This study is designed as cross-over double-blind placebo-controlled randomized clinical trial that 40 diabetic patients with sleep disorder with the inclusion criteria will enter into the study and randomly assign to first intervention and first placebo groups.The primary outcomes are change in sleep disorder and metabolic parameters that will be evaluated at the end of the study.

DETAILED DESCRIPTION:
Considering the high prevalence of sleep disturbance in diabetic patients and the effectiveness of lavender in treatment of sleep disorders in this study the efficacy of Lavender aromatherapy in sleep disorder and metabolic parameters in diabetic patients will be investigated. This study is designed as cross-over double-blind placebo-controlled randomized clinical trial that 40 diabetic patients with sleep disorder with the inclusion criteria will enter into the study and randomly assign to first intervention and first placebo groups.The primary outcomes are change in sleep disorder and metabolic parameters that will be evaluated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2
* Age between 25-65 years old
* Fasting Blood Sugar between 70-130
* 2 hour post prandial glucose less than 180.
* HbA1C less than 7
* Sleep disorder according to pittsburgh Insomnia Rating Scale more than 5.

Exclusion Criteria:

* Any systemic illnesses
* Use of sedative or antidepressant drugs
* Pregnancy
* Lactation
* History of allergic reaction to Lavender
* History of allergic rhinitis, asthma and respiratory disorders
* Anosmia
* Headache that start with smell
* Cigarette smocking or substance abuse
* Hospitalization or surgery within 1 months ago.
* Work shift

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Insomnia Rating Scale | 4 weeks
  evaluate the sleep disorder with Pittsburgh Insomnia Rating Scale

SECONDARY OUTCOMES:
Fasting Blood Sugar | 4 week
  blood sample
2 hours Post Prandial Glucose | 4 week
  blood sample
Serum Insulin | 4 week
  blood sample
C Reactive Protein | 4 week
  blood sample
Uric acid | 4 week
  blood sample
Creatinine | 4 week
  blood sample
Triglyceride | 4 week
  blood sample
Cholesterol | 4 week
  blood sample
Low Density Lipoprotein | 4 week
  blood sample
High Density Lipoprotein | 4 week
  blood sample
Aspartate Aminotransferase | 4 week
  blood sample
Alanine Aminotransferase | 4 week
  blood sample
weight | 4 week
  Scale
Body Mass Index | 4 week
  Body Mass Index
waist circumference | 4 week
  Meter
hip circumference | 4 week
  Meter
Systolic Blood Pressure | 4 week
  Blood Pressure measurement by digital sphygmometer
Diastolic Blood Pressure | 4 week
  Blood Pressure measurement by digital sphygmometer

CONTACTS AND LOCATIONS:
Overall Officials: Mesbah Shams, M.D., Study Chair — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences
Locations (2):
- Iran (2):
  - Shahid Motahhari Clinic, Shiraz University of Medical Sciences, Shiraz, Fars
  - Shiraz University of Medical Sciences, Shiraz, Fars